CLINICAL TRIAL: NCT02820753
Title: A Universal Medication Schedule to Promote Adherence to Complex Drug Regimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of North Carolina (Other); Emory University (Other); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Michael S. Wolf, Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01AG046352-01A1 (NIH)
Record Dates: First submitted 2016-05-16; First posted 2016-07-01 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Adherence
Keywords: Universal Medication Schedule; Health Literacy; Medication adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (No Intervention): Patients who have not received the initial 6 weeks of text message reminders telling them to take their medicines; or did not complete at least 1 portal survey that asks them if they filled their medications, if they had any side effects or concerns; or did not receive either intervention will be considered as enhanced usual care.
  Patients will only receive EHR tools (patient-friendly med-sheets about their medicines, MedList putting their medicines into the Universal Medication Schedule, and UMS sigs on their Rx bottles).
- Text or Portal (Active Comparator): Participants who received EHR strategies as well as, the initial 6 weeks of SMS messaging continuously that remind them to take their medicines; or logged on to the patient portal and completed at least one survey will be considered as receiving the intervention.
  Interventions: Behavioral: EHR + (Text or Portal)

INTERVENTIONS:
Behavioral: EHR + (Text or Portal) — Per protocol analysis:
  Patients who received the initial 6 weeks of SMS messaging continuously, or logged on to the patient portal and completed at least one survey.
  Arms: Text or Portal

SUMMARY:
This study will leverage available technologies and test strategies to impart the Universal Medication Schedule (UMS) in primary care to help patients understand, consolidate, safely use, and adhere to their complex medication regimens.

DETAILED DESCRIPTION:
The study investigators will conduct a patient-randomized controlled trial using a 2x2 factorial design to compare the effectiveness of interventions, alone or in combination, to one another. 1505 English and Spanish-speaking patients who are ≥ 50 years old, from a federally qualified health center (FQHC) in Chicago, and prescribed ≥ 3 Rx medications will be randomized to receive: 1) Enhanced Usual Care (EHR tools), 2) EHR tools + SMS, 3) EHR + Portal, or 4) EHR + SMS + Portal.

The study aims to:

1. Compare the effectiveness of the UMS EHR tools, with or without SMS and/or Portal interventions.
2. Evaluate the 'fidelity' (reliability) of each strategy and explore patient, staff, physician, and health system factors influencing the delivery of the interventions, alone and in combination
3. Assess the costs required to deliver each of the interventions from a health system perspective

Due to an NIA administrative hold, the interventions were not implemented as planned. Hence it was determined that the primary analysis would be "per-protocol" rather than intent-to-treat to assess the effect of the interventions under optimal conditions. Participants who either received the initial 6 weeks of SMS messaging continuously, or logged on to the patient portal and completed at least one survey will be considered as receiving the intervention. Those who have not received the initial 6 weeks of texting or completed at least 1 portal survey will be considered as enhanced usual care.

ELIGIBILITY:
Inclusion Criteria:

* age 50+
* English or Spanish speaking
* Prescribed 3+ medications
* Primarily responsible for administering own medication
* Owns a cell phone and feels comfortable receiving texts
* Access and proficient in using internet at home and has a personal email address

Exclusion Criteria:

* Major cognitive, visual, or hearing impairment
* Doesn't meet inclusion criteria.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Wolf, PHD, Principal Investigator — Northwestern University; Stacy C Bailey, PHD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bailey SC, Wismer GA, Parker RM, Walton SM, Wood AJJ, Wallia A, Brokenshire SA, Infanzon AC, Curtis LM, Kwasny MJ, Wolf MS. Development and rationale for a multifactorial, randomized controlled trial to test strategies to promote adherence to complex drug regimens among older adults. Contemp Clin Trials. 2017 Nov;62:21-26. doi: 10.1016/j.cct.2017.08.013. Epub 2017 Aug 18. PMID 28823927

RESULTS

PARTICIPANT FLOW:
Groups:
- Text or Portal: Participants who received EHR strategies as well as, the initial 6 weeks of SMS messaging continuously that remind them to take their medicines; or logged on to the patient portal and completed at least one survey will be considered as receiving the intervention.
  EHR + (Text or Portal): Per protocol analysis:
  Patients who received the initial 6 weeks of SMS messaging continuously, or logged on to the patient portal and completed at least one survey.
Period: Baseline
Arm/Group | Enhanced Usual Care | Text or Portal
Started | 256 | 421
Completed | 256 | 421
Not Completed | 0 | 0
Period: 2 Month
Arm/Group | Enhanced Usual Care | Text or Portal
Started | 256 | 421
Completed | 178 | 379
Not Completed | 78 | 42
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 24 | 26
Not completed — Stopped per NIH Hold | 51 | 13
Period: 6 Month
Arm/Group | Enhanced Usual Care | Text or Portal
Started | 253 | 418
Completed | 150 | 307
Not Completed | 103 | 111
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 20 | 27
Not completed — Stopped per NIH Hold | 81 | 81
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care | Text or Portal | Total
Number analyzed (Participants) | 256 | 421 | 677
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (6.4) | 61.0 (7.0) | 60.9 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 257 | 425
  Male | 88 | 164 | 252
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 5 | 11
  Asian | 6 | 8 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 60 | 96 | 156
  White | 174 | 294 | 468
  More than one race | 10 | 16 | 26
  Unknown or Not Reported | 0 | 2 | 2
Recruitment Site [Count of Participants; unit: Participants]
  Northwestern | 27 | 55 | 82
  Erie | 229 | 366 | 595
Health Literacy, Newest Vital Sign (NVS) [Count of Participants; unit: Participants]
  Limited | 109 | 151 | 260
  Marginal | 78 | 110 | 188
  Adequate | 68 | 160 | 228
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence - Pill Count
Description: Pill Count is conducted for all pill form medications using an electronic pill counter at baseline and 6 months. The proportion of pills taken over pills prescribed (PT/PP) will be calculated for each medication at each time point. Pills taken will be calculated by subtracting the number of pills from the total quantity prescribed. Pills prescribed will be calculated by multiplying the number of pills prescribed each day by the number of days since the medication was filled. A proportion of pills taken over pills prescribed (PT/PP) of 80% or more is considered adherent.
  Analyses were performed using 2-level Generalized linear models (PROC GENMOD), with medications nested in participants and with a logit link.
  Confounding variables, such as adherence at baseline, gender, age, language, health status and medication regimen complexity index (MRCI) were included as fixed effects in the models. Results are presented as predicted probabilities with 95% Confidence Intervals.
Time Frame: 6 months after Baseline
Population: Observations were excluded if: 1.Medications were not in pill form; 2.Participants couldn't provide quantities on their bottles; 3.Missing Fill or Start Dates, 4.Participants started their medications on the same date as their pill count date; 5. Missing medications labels; 6. Participants combined medication bottles and discarded their old bottles; 7. Pills taken > Quantity on bottle; 8. PRN Medications
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability of adherence (PT/PP => 0.8)
Units Other Than Participants: Medications
Arm/Group | Enhanced Usual Care | Text or Portal
Number analyzed (Participants) | 143 | 293
Number analyzed (Medications) | 559 | 1189
Probability of adherence (PT/PP => 0.8) | 0.46 [0.41 to 0.52] | 0.53 [0.48 to 0.57]
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Text or Portal; Test type: Superiority; p = 0.04, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; Mean Difference (Net) = 0.26, 95% CI 2-sided [0.01 to 0.51] — Treatment difference = (Text or Portal) - Enhanced Usual Care

2. Primary Outcome: Medication Adherence - Proper Use
Description: Participants are asked questions about their 24 hour recall of medication use for each of their medications; they are asked to specify the amount taken (dose), the number of times the med was taken (frequency), the total number of pills taken, and when the doses were taken (to calculate spacing: hours between doses). Proper Use will be scored as yes or no, reflecting having demonstrated all of the following: correct dose, frequency, total and spacing based on the medication bottle instructions. Results are presented as predicted probabilities with 95% Confidence Intervals.
  Analyses were performed using 2-level Generalized linear models (PROC GENMOD), with medications nested in participants and with a logit link.
  Confounding variables, such as recruitment time, clinic, health status, gender, age, time effect, and medication regimen complexity index (MRCI) were included as fixed effects in the models.
Time Frame: 6 Months after Baseline
Population: Observations were excluded if 1. the medication bottle had a missing label, or 2. participants did not complete the 24 hour med recall use questions
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability of Proper Use (Yes)
Units Other Than Participants: Medications
Arm/Group | Enhanced Usual Care | Text or Portal
Number analyzed (Participants) | 255 | 421
Number analyzed (Medications) | 5854 | 11208
Probability of Proper Use (Yes) | 0.71 [0.68 to 0.73] | 0.71 [0.69 to 0.73]
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Text or Portal; Test type: Superiority; p = 0.53, Mixed Models Analysis — The threshold for statistical significance was p < 0.05; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.08 to 0.15] — Treatment Difference = (Text or Portal - Enhanced Usual Care

3. Primary Outcome: Medication Adherence - ASK12
Description: Participants completed the ASK-12 questionnaire, a brief measure of adherence that cover three key domains: inconvenience/forgetfulness, treatment beliefs and behavior.
  The ASK-12 is scored by summing the selected responses (with scores ranging from 12 to 60) with higher scores indicating greater barriers to adherence.
  Analyses were performed using Generalized linear models (PROC GENMOD), with a repeated subject effect, and an identity link.
  Confounding variables such as health status, gender, age, health activation (CHAI), language, time effect and number of chronic conditions were included as fixed effects in the models. Results are presented as predicted probabilities with 95% Confidence Intervals.
Time Frame: 6 Months after Baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Enhanced Usual Care | Text or Portal
Number analyzed (Participants) | 255 | 421
score on a scale | 22.40 [21.75 to 23.05] | 22.06 [21.48 to 22.65]
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Text or Portal; Test type: Superiority; p = 0.41, Mixed Models Analysis — The threshold for significance is p < 0.05; Mean Difference (Net) = -0.34, 95% CI 2-sided [-1.16 to 0.48] — Treatment Difference = (Text or Portal) - Enhanced Usual Care

4. Other Pre Specified Outcome: Systolic Blood Pressure
Description: Systolic blood pressure will be collected on all participants at baseline and 6 months.
  Change of Systolic blood pressure from baseline will be measured, only in those who are diagnosed with hypertension. Negative Least Square Means indicate a decrease of systolic blood pressure, whereas a positive Least Square Means indicate an increase of systolic blood pressure by 6 Months.
  Analyses were performed using Generalized linear models (PROC GENMOD), with an identity link.
  Confounding variables, such as mean systolic blood pressure at baseline, gender, age, race, and number of prescribed medications were included as fixed effects in the models. Results are presented as adjusted least square means with 95% Confidence Intervals.
Time Frame: 6 months after Baseline
Population: This measure was only used for participants who are diagnosed with hypertension, those who are not were not included.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Enhanced Usual Care | Text or Portal
Number analyzed (Participants) | 147 | 260
mmHg | -0.04 [-3.73 to 3.64] | 1.79 [-1.60 to 5.18]
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Text or Portal; Test type: Superiority; p = 0.27, Mixed Models Analysis — The threshold for significance is p < 0.05; Mean Difference (Net) = 1.83, 95% CI 2-sided [-1.39 to 5.06] — Treatment difference = (Text or Portal ) - Enhanced Usual Care

5. Other Pre Specified Outcome: Hemoglobin A1c
Description: Hemoglobin A1c (hbA1c) will be collected on diabetic patients only, at baseline and 6 months.
  Change of hbA1c from baseline is modelled. A positive Least Square Mean indicates an increase of hbA1c at 6 months, whereas a negative Least Square Mean indicates a decrease of hbA1c.
  Analyses were performed using Generalized linear models (PROC GENMOD), with an identity link.
  Confounding variables, such as hbA1c at baseline, gender, age, health status, language, medication regimen complexity index (MRCI), and health literacy (Newest Vital Sign) were included as fixed effects in the models. Results are presented as adjusted least square means with 95% Confidence Intervals.
Time Frame: 6 months after Baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | Enhanced Usual Care | Text or Portal
Number analyzed (Participants) | 56 | 115
percentage of glycated hemoglobin | 0.23 [-0.18 to 0.64] | 0.003 [-0.28 to 0.29]
Statistical Analysis 1: Comparison: Enhanced Usual Care; Test type: Superiority; p = 0.33, Mixed Models Analysis — The threshold for significance is p < 0.05; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.68 to 0.23] — Treatment Difference = (Text or Portal) - Enhanced Usual Care

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Enhanced Usual Care | Text or Portal
All-Cause Mortality (participants affected / at risk) | 0/256 | 1/421
Serious Adverse Events (participants affected / at risk) | 0/256 | 0/421
Other Adverse Events (participants affected / at risk) | 0/256 | 0/421

LIMITATIONS AND CAVEATS:
Due to an NIA administrative hold from July 2018-April 2019, recruitment has halted for that time period and the interventions were not implemented as planned. Hence it was determined that the primary analysis would be "per-protocol" rather than intent-to-treat to assess the effect of the interventions under optimal conditions. Additionally, due to restrictions to in-person interviews due to COVID-19, we were unable to recruit new patients starting March 12, 2020

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT02820753/Prot_SAP_000.pdf